CLINICAL TRIAL: NCT03081195
Title: SMART Africa: Addressing African Youth Mental Health by Scaling Family and Community-Level EBPs
Brief Title: SMART Africa (Strengthening Mental Health Research and Training)
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Ghana (Other); University of Nairobi (Other); Reach the Youth Uganda (Other); New York University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19MH110001-011; U19MH110001 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-16 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Comparison Group; Multiple Family Groups by Parent Peers; Multiple Family Groups by Community Health Workers
Keywords: child behavior; intervention; multiple family group; Sub Saharan Africa; caregivers
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Schools will be randomly assigned to 3 study conditions: 1) MFG-delivered by trained family peers; 2) MFG-delivered by community health workers; or, 3) Comparison: Mental health and school support materials (books).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MFG-delivered by trained family peers (Experimental): MFG delivered by trained parent peers drawn from local school planning councils:
  10 schools; 60 parent peers (6 per school x 10); 1,000 children and adult caregivers; children screened to evidence serious emerging and clinically significant DBDs
  Interventions: Behavioral: MFG
- MFG-delivered by CHWs (Experimental): MFG delivered by community health workers (CHW) drawn from local primary care clinics:
  10 schools; 60 community health workers (6 assigned to children per school x 10); 1,000 children and adult caregivers; children screened to evidence serious emerging and clinically significant DBDs
  Interventions: Behavioral: MFG
- Bolstered care (No Intervention): Comparison (Bolstered care): Mental health wellness materials and educational supports (e.g. books, uniforms)
  10 schools; 1,000 children and adult caregivers; children screened to evidence serious emerging and clinically significant DBDs

INTERVENTIONS:
Behavioral: MFG — The MFG is a series of weekly meetings guided by a protocol.Over the course of 16 weeks, groups are held weekly and are facilitated by trained and supervised group leaders (in this case either parent peers or community health outreach workers). Groups can consist of up to 20 families involving adult caregivers and all children over six years of age in the family. The protocols have been designed to provide opportunities during each session to directly apply content to the realities of family life, emergent cultural and values perspectives, as well as tailor messages to age of child. Redundancy for missed appointments and opportunities for reinforcement is built in. We aim for families to attend at least 8 meetings or more (out of 16 sessions in total), as findings suggests this dose is needed to reduce child conduct problems and the majority of families reach this goal.
  Other Names: 4Rs and 2Ss; Amaka Amasanyufu (Happy Families in Luganda-Uganda); Dang-Malgu (Family Togetherness in Dagbani-Ghana)
  Arms: MFG-delivered by CHWs; MFG-delivered by trained family peers

SUMMARY:
The objective of this research study is to examine the implementation of and outcomes associated with an evidence-based practice (EBP), specifically Multiple Family Group (MFG) targeting youth disruptive behavior challenges and success, through a scale up intervention study in Uganda, and two pilot studies that will be conducted in Kenya and Ghana.

DETAILED DESCRIPTION:
A longitudinal experimental mixed methods effectiveness-implementation hybrid research design will be employed. The study will be conducted across thirty primary schools representing both semi-urban and rural communities. We expect to involve 3,000 youth (in primary schools grades 2 through 7; 8 to 13 years) and their adult caregivers (3,000) in Uganda, 180 youth and their caregivers (180) in Ghana, and 180 youth and their caregivers (180) in Kenya.

Schools will be randomly assigned to 3 study conditions: 1) MFG-delivered by trained family peers; 2) MFG-delivered by community health workers (school health education program coordinators in Ghana); or, 3) Comparison: mental health and school support materials (e.g., books, uniforms). Data will be collected at baseline, 8 and 16 weeks, and 6 months follow-up (10 months from baseline).

More specifically the objectives of this study are:

Primary objectives

1. To examine short- and long-term outcomes associated with the MFG. Hypothesis: Children in the treatment groups (MFG) will improve significantly more compared to those in the comparison (usual care) group.
2. To examine how systematic variations in the delivery of an evidence-based MFG program impacts outcomes for children with behavioral difficulties and their caregivers in each country context.

   Hypothesis: Children who participate in MFG with their families will display significantly reduced conduct difficulties and increased functioning over time compared to those involved in comparison condition. We expect that parent peers - compared to community health workers - will evidence significantly more success engaging families to attend MFG sessions, thus, children in the MFG-parent peer delivered condition will evidence the great improvement relative to the other two study conditions.

   Secondary objectives
3. To compare the uptake and implementation of MFGs by trained existing family peers and community outreach health workers.

   Hypothesis: Given the level of training that community outreach health workers have received prior to the study as part of their regular professional training, they will evidence higher fidelity initially, yet with training and ongoing supervision, we expect these differences to decrease over time.
4. To examine multi-level (state/government, NGOs, families, schools, communities) influences on the uptake, implementation, effectiveness and sustainability of EBPs that address serious child disruptive behavioral challenges.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria for caregiver/child dyads:

* Adult caregiver of a child in primary school, grades two through 7, ages 8 to 13 years
* Adult caregiver willing to consent and available for research and intervention activities
* Child between the ages 8 to 13 or in primary school (grades two through seven) who is screened for ODD or CD as measured by the Disruptive Behavior Disorder Rating Scale, Impairment Scale, and Iowa Conners Scale.
* Child willing to assent.

  * Inclusion criteria for parent peers:
* Caregivers of children who agree to be trained to provide support to families.

  * Inclusion criteria for community health workers
* Lay paraprofessionals who work within primary care settings.

  * Inclusion criteria for school directors
* Directors who oversee schools where the proposed intervention will have been tested.

Exclusion Criteria:

- Exclusion criteria for caregiver/child dyads:

* Lack of understanding of study and study procedures as determined by the research team
* Child or caregiver refusal to participate

  * Exclusion criteria for parent peers:
* Refusal to participate

  * Exclusion criteria for community health workers
* Refusal to participate

  * Exclusion criteria for school directors
* Refusal to participate

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3117 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Child disruptive behavior | baseline, 8 weeks, 16 weeks, 6 months
  Change in disruptive behavior will be measured by Iowa Connors
Child impairment | baseline, 8 weeks, 16 weeks, 6 months
  Change in disruptive behavior will be measured Impairment scale

SECONDARY OUTCOMES:
Implementation and Feasibility | 8 weeks, 16 weeks, 6 months
  implementation and feasibility checklist measures
Fidelity | end of session at week 1, week 2, week 3, week 4, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14, week 15, week 16
  MFG Intervention Fidelity Assessment measures
Sustainability | 8 weeks, 16 weeks, 6 months
  Program Sustainability Assessment Tool
Implementation process | 8 weeks, 16 weeks, 6 months
  Metropolitan Area Child Study process measure
Parenting | baseline, 8 weeks, 16 weeks, 6 months
  Change in parenting will be measured by Alabama Parenting questionnaire
Social support | baseline, 8 weeks, 16 weeks, 6 months
  Improvement in social support will be measured by Multidimensional scale of perceived social support -modified
Caregiver depression | baseline, 8 weeks, 16 weeks, 6 months
  Change in caregiver depression will be measured by Center for Epidemiologic Studies Short Depression Scale
Caregiver mental health | baseline, 8 weeks, 16 weeks, 6 months
  Change in caregiver mental health will be measured by Brief Symptom Checklist
Caregiver stress | baseline, 8 weeks, 16 weeks, 6 months
  Change in caregiver stress will be measured by parent stress index short form
Child mental health | baseline, 8 weeks, 16 weeks, 6 months
  Change in Child mental health will be measured by Strengths and Difficulties questionnaire
Child self-concept | baseline, 8 weeks, 16 weeks, 6 months
  Change in child self-concept will be measured by tennessee self-concept
Child depression | baseline, 8 weeks, 16 weeks, 6 months
  Change in child depression will be measured by child depression scale
Family relations | baseline, 8 weeks, 16 weeks, 6 months
  Change in family relations will be measured by Family Relations and Cohesion scale

CONTACTS AND LOCATIONS:
Overall Officials: Mary McKay, PhD, Principal Investigator — Washington University School of Medicine; Fred Ssewamala, PhD, Principal Investigator — Washington University School of Medicine
Locations (4):
- Washington University in St. Louis, St Louis, Missouri, United States
- University of Ghana, Accra, Ghana
- University of Nairobi, Nairobi, Kenya
- Reach the Youth Uganda, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: No
There will be no individual participant data that will be shared.

REFERENCES:
- [Derived] Ssewamala FM, Brathwaite R, Sensoy Bahar O, Namatovu P, Neilands TB, Kiyingi J, Huang KY, McKay MM. The Post-intervention Impact of Amaka Amasanyufu on Behavioral and Mental Health Functioning of Children and Adolescents in Low-Resource Communities in Uganda: Analysis of a Cluster-Randomized Trial From the SMART Africa-Uganda Study (2016-2022). J Adolesc Health. 2023 May;72(5S):S3-S10. doi: 10.1016/j.jadohealth.2022.09.035. PMID 37062581
- [Derived] Brathwaite R, Sensoy Bahar O, Mutumba M, Byansi W, Namatovu P, Namuwonge F, Neilands TB, McKay MM, Hoagwood KE, Ssewamala FM. Short-Term Impact of "Amaka Amasanyufu" Multiple Family Group Intervention on Mental Health Functioning of Children With Disruptive Behavior Disorders in Uganda. J Am Acad Child Adolesc Psychiatry. 2023 Jul;62(7):777-790. doi: 10.1016/j.jaac.2022.12.028. Epub 2023 Mar 8. PMID 36898607
- [Derived] Brathwaite R, Ssewamala FM, Sensoy Bahar O, McKay MM, Neilands TB, Namatovu P, Kiyingi J, Zmachinski L, Nabayinda J, Huang KY, Kivumbi A, Bhana A, Mwebembezi A, Petersen I, Hoagwood K; SMART Africa - Uganda Field Team. The longitudinal impact of an evidence-based multiple family group intervention (Amaka Amasanyufu) on oppositional defiant disorder and impaired functioning among children in Uganda: analysis of a cluster randomized trial from the SMART Africa-Uganda scale-up study (2016-2022). J Child Psychol Psychiatry. 2022 Nov;63(11):1252-1260. doi: 10.1111/jcpp.13566. Epub 2022 Jan 6. PMID 34989404
- [Derived] Asampong E, Ibrahim A, Sensoy-Bahar O, Kumbelim K, Yaro PB, McKay MM, Ssewamala FM. Adaptation and Implementation of the Multiple-Family Group Intervention in Ghana. Psychiatr Serv. 2021 May 1;72(5):571-577. doi: 10.1176/appi.ps.201900626. Epub 2021 Jan 12. PMID 33430647
- [Derived] Ssewamala FM, Sensoy Bahar O, McKay MM, Hoagwood K, Huang KY, Pringle B. Strengthening mental health and research training in Sub-Saharan Africa (SMART Africa): Uganda study protocol. Trials. 2018 Aug 6;19(1):423. doi: 10.1186/s13063-018-2751-z. PMID 30081967